CLINICAL TRIAL: NCT05325775
Title: A Phase 2A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy, Safety and Pharmacokinetics (PK) of ACER-801 for Treatment of Moderate to Severe Vasomotor Symptoms (VMS) Associated With Menopause
Brief Title: Dose-ranging, PK, Safety, Efficacy Study of Osanetant in Patients With Moderate/Severe VMS Associated With Menopause
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acer Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACER-801-201
Record Dates: First submitted 2022-03-27; First posted 2022-04-13 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-06

CONDITIONS: Post-menopausal Vasomotor Symptoms
MeSH Terms: interventions — BID protein, human; SR 142801

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1:1:1 ratio to ACER-801 per one of the following dosing schedules prior to dosing:
  * 50 mg BID,
  * 100 mg BID,
  * 200 mg BID, or
  * Placebo BID
  Each arm is administered orally for 14 consecutive days (28 doses).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, the Investigator, and other members of the staff involved with the study will remain blinded to study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ACER-801 50 mg BID (Experimental): ACER-801 (osanetant) 50 mg BID (1 x 50 mg and 3 x placebo, twice daily)
  Interventions: Drug: ACER-801 50 mg BID
- ACER-801 100 mg BID (Experimental): ACER-801 (osanetant) 100 mg BID (2 x 50 mg and 2 x placebo, twice daily)
  Interventions: Drug: ACER-801 100 mg BID
- ACER-801 200 mg BID (Experimental): ACER-801 (osanetant) 200 mg BID (4 x 50 mg and 0 x placebo, twice daily)
  Interventions: Drug: ACER-801 200 mg BID
- Placebo (Placebo Comparator): Placebo (4 x Placebo of ACER-801 twice daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACER-801 50 mg BID — 50 mg BID (twice daily)
  Other Names: osanetant
  Arms: ACER-801 50 mg BID
Drug: ACER-801 100 mg BID — 100 mg BID (twice daily)
  Other Names: osanetant
  Arms: ACER-801 100 mg BID
Drug: ACER-801 200 mg BID — 200 mg BID (twice daily)
  Other Names: osanetant
  Arms: ACER-801 200 mg BID
Drug: Placebo — Placebo
  Other Names: Placebo of ACER-801
  Arms: Placebo

SUMMARY:
In this clinical research study, subjects will be given the study drug, ACER-801 (osanetant) or placebo (looks like the study drug but contains no active ingredients). The study drug works on a receptor in the brain and the intended purpose is for the study treatment of moderate to severe Vasomotor Symptoms (VMS) also referred to as hot flashes or flushes associated with menopause. Hot flashes are a change in your temperature that occurs due to changes in your hormones.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled, dose-ranging study in post menopausal women in which the pharmacokinetics, safety and efficacy of ACER-801 (osanetant 50 mg twice daily [BID], 100 mg BID, and 200 mg BID) will be compared to placebo.

Subjects will enter a Screening Period to determine eligibility. Subjects will be required to complete hot flash diaries for 2 weeks prior to randomization. Eligible subjects will be admitted to a Clinical Research Unit and remain in the clinic for 14 days after completion of treatment and all study assessments. The study includes a 14 day safety follow-up assessment. Subjects will be randomized in a 1:1:1:1 ratio.

ELIGIBILITY:
Key Inclusion Criteria:

1. Post-menopausal female subjects 40-65 years of age, inclusive.

   Menopause will be defined as:
   1. At least 12 months of spontaneous, continuous amenorrhea, or
   2. At least 6 months of spontaneous, continuous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/mL at screening, or
   3. At least 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
2. At baseline women:

   1. With an average number of moderate to severe hot flashes/day for 2 weeks prior to randomization (per continuous hot flash diary).
   2. That have a change of < 50% in average 24-hour hot flash frequency 2 weeks prior to randomization.

      * Moderate: defined as sensation of heat with sweating, able to continue activity.
      * Severe: defined as sensation of heat with sweating, causing cessation of activity.

Key Exclusion Criteria:

1. Any active comorbid disease deemed by the investigator to be clinically significant, which could impact safety during study conduct including renal or hepatic impairment.
2. Use of any prohibited medications.
3. Body mass index (BMI) >35 kg/m2.
4. Any active ongoing condition that could cause difficulty in interpreting vasomotor symptoms.
5. Inability to complete questionnaires and continuous hot flash diary for any reason.
6. Subjects who, in the opinion of the investigator, should not participate in the study for any other reason.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Boston, MSN, APNP, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Started | 12 | 12 | 12 | 13
Completed | 12 | 12 | 12 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Post menopausal women 40-65 years of age, inclusive
Groups:
- Total: Total of all reporting groups
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 13 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 13 | 49
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (4.25) | 55.6 (5.58) | 57.3 (5.31) | 56.5 (3.31) | 56.2 (4.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 12 | 13 | 49
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 7 | 5 | 18
  Not Hispanic or Latino | 8 | 10 | 5 | 8 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 2 | 1 | 12
  White | 8 | 7 | 9 | 11 | 35
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 13 | 49
Frequency of vasomotor symptoms [Mean (Standard Deviation); unit: daily number of symptoms] — Baseline frequency was calculated by totaling the number of mild, moderate and severe hot flashes reported during the baseline period (Days -14 to -1, inclusive).
  All denominators were adjusted to account for the actual number of baseline period days data was collected.
  daily number of symptoms | 11.77 (1.898) | 13.05 (3.748) | 11.58 (1.932) | 13.42 (3.215) | 12.46 (2.70)
Severity of vasomotor symptoms / hot flash severity [Mean (Standard Deviation); unit: score on a scale] — Baseline severity was calculated for each subject using the following formula: [(1 × number of mild hot flashes) + (2 × number of moderate hot flashes) + (3 × number of severe hot flashes)]/total number of hot flashes reported. Baseline was defined as the average severity value calculated using data collected during the baseline period (Days -14 to -1, inclusive).
  Severity scale ranges from 1 (mild) to 3 (severe). All denominators were adjusted to account for the actual number of baseline period days data was collected.
  score on a scale | 2.28 (0.204) | 2.36 (0.156) | 2.28 (0.255) | 2.39 (0.247) | 2.33 (0.216)
Hot Flash Severity Score [Mean (Standard Deviation); unit: score on a scale] — The hot flash severity score is a composite of the frequency and severity of hot flashes, and was calculated as follows: [number of mild hot flashes on Day Y x 1] + [number of moderate hot flashes on Day Y x 2] + [number of severe hot flashes on Day Y x 3].
  Baseline period is defined as the average severity score using data collected from Days-14 to -1, inclusive. Denominators were adjusted to account for the actual number of days data was collected.
  score on a scale | 26.89 (4.388) | 30.43 (8.122) | 26.35 (4.797) | 31.86 (7.848) | 28.88 (6.289)

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax) of ACER-801
Description: maximum concentration of ACER-801 measured at Day 1
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only Cmax (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 1
Population: All subjects in the safety population who have sufficient plasma concentration above the limit of quantitation. PK is not tested in placebo arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 10.78 (8.97) | 32.36 (33.56) | 41.75 (30.69)

2. Primary Outcome: Peak Plasma Concentration (Cmax) of ACER-801
Description: maximum concentration of ACER-801 measured at Day 14
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only Cmax (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 27.47 (22.09) | 83.08 (52.38) | 168.28 (89.68)

3. Primary Outcome: Peak Plasma Concentration (Cmax) of ACER-801 Metabolite
Description: peak concentration of ACER-801 metabolite measured at Day 1
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only Cmax (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 15.25 (11.60) | 43.77 (44.58) | 61.31 (38.44)

4. Primary Outcome: Peak Plasma Concentration (Cmax) of ACER-801 Metabolite
Description: peak concentration of ACER-801 metabolite measured at Day 14
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only Cmax (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 38.79 (27.56) | 92.17 (52.18) | 196.80 (92.74)

5. Primary Outcome: Time to Reach Maximum Concentration (Tmax) of ACER-801
Description: time to reach maximum concentration of ACER-801 measured at Day 1
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only Tmax (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
hour | 1.29 (0.66) | 1.21 (0.54) | 1.33 (0.58)

6. Primary Outcome: Time to Reach Maximum Concentration (Tmax) of ACER-801
Description: time to reach maximum concentration of ACER-801 at Day 14
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only Tmax (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
hour | 0.96 (0.33) | 2.17 (1.45) | 1.79 (0.75)

7. Primary Outcome: Time to Reach Maximum Concentration (Tmax) of ACER-801 Metabolite
Description: time to reach maximum concentration of ACER-801 metabolite at Day 1
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only Tmax (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
hour | 1.38 (0.53) | 1.25 (0.54) | 1.33 (0.54)

8. Primary Outcome: Time to Reach Maximum Concentration (Tmax) of ACER-801 Metabolite
Description: Time to reach maximum concentration of ACER-801 metabolite at Day 14
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only Tmax (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
hour | 1.21 (0.45) | 2.21 (0.92) | 1.88 (0.61)

9. Primary Outcome: Area Under the Concentration Curve From Dosing to the Time of the Last Measured Concentration (AUClast) of ACER-801
Description: Area under the concentration time curve (AUC) from the time of dosing (0 hour) to the time of the last quantifiable (positive) concentration (Tlast) of ACER-801, calculated by a combination of linear and logarithmic trapezoidal methods (linear up/log down method)
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only AUClast (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 42.32 (37.02) | 149.92 (159.83) | 205.94 (156.95)

10. Primary Outcome: Area Under the Concentration Curve From Dosing to the Time of the Last Measured Concentration (AUClast) of ACER-801
Description: as for outcome 9
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 174.72 (150.61) | 517.91 (346.91) | 1252.54 (769.07)

11. Primary Outcome: Area Under the Concentration Curve From Dosing to the Time of the Last Measured Concentration (AUClast) of ACER-801 Metabolite
Description: Area under the concentration time curve (AUC) from the time of dosing (0 hour) to the time of the last quantifiable (positive) concentration (Tlast) of ACER-801 metabolite, calculated by a combination of linear and logarithmic trapezoidal methods (linear up/log down method)
  Blood sampling included predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 hrs (prior to evening dose) and 15 hrs post morning dose. Only AUClast (mean, SD) data are available due to abbreviated data analyses.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 61.42 (46.41) | 172.18 (165.54) | 291.23 (203.43)

12. Primary Outcome: Area Under the Concentration Curve From Dosing to the Time of the Last Measured Concentration (AUClast) of ACER-801 Metabolite
Description: as for outcome 11
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 257.56 (200.63) | 628.87 (383.91) | 1579.25 (847.47)

13. Primary Outcome: Half-life (T1/2) of ACER-801
Description: Terminal elimination half-life of ACER-801
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
hour | 5.17 (1.39) | 4.61 (1.26) | 4.80 (0.74)

14. Primary Outcome: Half-life (T1/2) of ACER-801
Description: Terminal elimination half-life of ACER-801
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
hour | 5.75 (1.05) | 5.06 (0.97) | 5.56 (1.15)

15. Primary Outcome: Half-life (T1/2) of ACER-801 Metabolite
Description: Terminal elimination half-life of ACER-801 metabolite
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
hour | 4.83 (1.30) | 4.83 (1.05) | 4.61 (0.66)

16. Primary Outcome: Half-life (T1/2) of ACER-801 Metabolite
Description: Terminal elimination half-life of ACER-801 metabolite
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
hour | 6.55 (1.41) | 5.57 (1.13) | 5.99 (1.55)

17. Primary Outcome: Number and Percentage of Adverse Events ≥ 5%
Description: An Adverse Event (AE) is defined as any untoward medical occurrence associated with the use of the investigational product in humans, whether or not considered related to investigational product. An AE can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with any use of the investigational product, without any judgment about causality and irrespective of route of administration, formulation, or dose, including an overdose.
Time Frame: 2 weeks
Population: Safety Population
Measure: Number; unit: events
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
events | 17 | 21 | 23 | 21

18. Primary Outcome: Number and Percentage of Serious Adverse Events (SAE)
Description: An AE is considered "serious" if, in the view of either the investigator or Acer, it results in any of the following outcomes: Death, Is immediately life threatening; Requires in-patient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability or incapacity; Results in a congenital abnormality or birth defect; Is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above.
Time Frame: 2 weeks
Population: Safety population
Measure: Number; unit: event(s)
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
event(s) | 0 | 0 | 1 | 0

19. Primary Outcome: Number and Percentage of Subjects Who Discontinued From the Study
Description: Discontinuation or withdrawal from the study.
Time Frame: Over 2 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
participants | 0 | 0 | 0 | 0

20. Primary Outcome: Number of Patients With a Clinically Significant Change From Baseline in Abnormalities Detected During Physical Examination
Description: A physician or appropriately qualified delegate conducted a full physical examination at baseline and at Day 14. The investigator decides if findings are considered abnormal at baseline and at Day 14 and whether the change is clinically significant. Only clinically significant changes will be reported.
Time Frame: At Day 14 relative to Baseline
Population: Safety Population
Measure: Number; unit: patients
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
patients | 0 | 0 | 0 | 0

21. Primary Outcome: Accumulation Ratio for Cmax (ARcmax) of ACER-801
Description: Cmax (maximum concentration) Accumulation Ratio calculated as Cmax,Day14/ Cmax,Day1 and AUCt,Day14/ AUCt,Day1, where the dosing interval t is 12h.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ratio | 4.87 (6.36) | 4.38 (4.69) | 4.76 (1.78)

22. Primary Outcome: Accumulation Ratio for AUC (ARauc) of ACER-801
Description: AUC (area under the curve) Accumulation Ratio calculated as Cmax,Day14/ Cmax,Day1 and AUCt,Day14/ AUCt,Day1, where the dosing interval t is 12h.
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ratio | 7.76 (8.33) | 6.15 (6.85) | 7.16 (2.46)

23. Primary Outcome: Accumulation Ratio for Cmax (ARcmax) of ACER-801 Metabolite
Description: as for outcome 21
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ratio | 4.28 (4.76) | 2.70 (1.48) | 3.51 (1.29)

24. Primary Outcome: Accumulation Ratio for AUC (ARauc) of ACER-801 Metabolite
Description: as for outcome 22
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ratio | 5.99 (5.58) | 5.11 (4.14) | 6.22 (2.26)

25. Primary Outcome: Metabolite: Parent Ratio of AUC (MRauc)
Description: MR = Metabolite:Parent Ratio calculated as Cm,day14/ Cp,day1 and AUCt,m,day14/ AUCt,p,day1, where m and p are the metabolite and parent drug, respectively, and t is the dosing interval (12 h).
  AUC = area under the curve
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ratio | 1.97 (1.33) | 1.34 (0.34) | 1.53 (0.33)

26. Primary Outcome: Metabolite: Parent Ratio of AUC (MRauc)
Description: AUC (area under the curve) MR = Metabolite:Parent Ratio calculated as Cm,day14/ Cp,day1 and AUCt,m,day14/ AUCt,p,day1, where m and p are the metabolite and parent drug, respectively, and t is the dosing interval (12 h).
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ratio | 1.65 (0.30) | 1.23 (0.18) | 1.31 (0.13)

27. Primary Outcome: Metabolite:Parent Ratio of Cmax (MRcmax)
Description: MR = Metabolite:Parent Ratio calculated as Cm,day14/ Cp,day1 and AUCt,m,day14/ AUCt,p,day1, where m and p are the metabolite and parent drug, respectively, and t is the dosing interval (12 h).
  ACER-801 (parent); Cmax (maximum concentration)
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ratio | 1.55 (0.24) | 1.61 (0.60) | 1.69 (0.58)

28. Primary Outcome: Metabolite:Parent Ratio of Cmax (MRcmax)
Description: as for outcome 27
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
ratio | 1.55 (0.24) | 1.15 (0.19) | 1.23 (0.17)

29. Primary Outcome: Area Under the Concentration Curve From t0 to Infinite Time (AUCinf) of ACER-801
Description: AUC from the time of dosing (0 hour) extrapolated to infinity, calculated as AUClast + Clast/λz, where Clast was the last quantifiable concentration, and λz was the terminal elimination rate constant Reliability of AUCinf values was contingent upon AUCext and λz Profiles with AUCext ≤20% and a λz which met reporting criteria were considered reliable and AUCinf was reported. For profiles that did not meet these criteria, AUCinf and any parameter requiring AUCinf for computation were not reported.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 53.50 (48.08) | 173.72 (178.05) | 247.19 (181.87)

30. Primary Outcome: Area Under the Concentration Curve From t0 to Infinite Time (AUCinf) of ACER-801
Description: as for outcome 29
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 231.48 (202.58) | 682.25 (393.98) | 1673.06 (1146.58)

31. Primary Outcome: Area Under the Concentration Curve From t0 to Infinite Time (AUCinf) of ACER-801 Metabolite
Description: as for outcome 29
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 76.92 (61.90) | 206.14 (193.55) | 347.35 (245.92)

32. Primary Outcome: Area Under the Concentration Curve From t0 to Infinite Time (AUCinf) of ACER-801 Metabolite
Description: as for outcome 29
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 380.43 (325.41) | 819.29 (496.58) | 2270.60 (1568.80)

33. Primary Outcome: Number of Subjects With a Clinically Significant Change From Baseline for Clinical Laboratory Evaluations: HEMATOLOGY
Description: Blood samples will be measured for hemoglobin, hematocrit, white blood count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), platelet count, red blood cell count (including mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration). Only clinically significant changes will be reported.
Time Frame: Over 2 weeks
Population: Safety population; transient changes from normal to low or high values were reported but none were deemed clinically significant.
Measure: Number; unit: participants
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
participants | 0 | 0 | 0 | 0

34. Primary Outcome: Number of Subjects With a Clinically Significant Change From Baseline for Clinical Laboratory Evaluations: SERUM CHEMISTRY
Description: Blood samples will be measured for albumin, alkaline phosphatase, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen, calcium, carbon dioxide, chloride, potassium, sodium, total cholesterol, creatinine, gamma glutamyl transferase, glucose, lactate dehydrogenase, phosphorus, total protein, uric acid. Only clinically significant changes will be reported.
Time Frame: 2 weeks
Population: as for outcome 33
Measure: Number; unit: participants
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
participants | 0 | 0 | 0 | 0

35. Primary Outcome: Number of Subjects With a Clinically Significant Change From Baseline for Clinical Laboratory Evaluations: COAGULATION
Description: Blood samples will be measured for prothrombin time, partial thromboplastin time, international normalized ratio. Only clinically significant changes will be reported.
Time Frame: 2 weeks
Population: as for outcome 33
Measure: Number; unit: participants
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
participants | 0 | 0 | 0 | 0

36. Primary Outcome: Number of Subjects With a Clinically Significant Change From Baseline for Clinical Laboratory Evaluations: URINALYSIS
Description: Urine samples will be measured for pH, specific gravity, protein, glucose, ketones, bilirubin. Only clinically significant changes will be reported.
Time Frame: 2 weeks
Population: as for outcome 33
Measure: Number; unit: participants
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
participants | 0 | 0 | 0 | 0

37. Primary Outcome: Number of Subjects With a Clinically Significant Change From Baseline for Clinical Laboratory Evaluations: BONE DENSITY MARKERS
Description: Blood samples not available/collected for testing. Blood samples will be measured for Bone Specific Alkaline Phosphatase (BSAP), osteocalcin, amino terminal propeptide of type 1 collagen (P1NP) and Collagen Type- C-Telopeptide (CTX). Only clinically significant changes will be reported.
Time Frame: 2 weeks
Population: Safety population. Hormone testing was not conducted. Blood samples not available/collected for testing.
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

38. Primary Outcome: Number of Subjects With a Clinically Significant Change From Baseline for Clinical Laboratory Evaluations: HORMONES
Description: Blood samples not available/collected for testing. Blood samples will be measured for catecholamines, vasopressin, gonadotropins, estradiol, testosterone, follicle stimulating hormone (FSH), luteinizing hormone (LH), adrenocorticotropic hormone (ACTH), cortisol, thyroid-stimulating hormone (TSH), T3 (Total and Free), T4 (Total and Free), prolactin, sex hormone binding globulin (SHBG), and insulin. Only clinically significant changes will be reported.
Time Frame: 2 weeks
Population: Safety population. Hormone testing was not conducted. Blood samples not available/collected for testing.
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

39. Secondary Outcome: Change in Frequency of Vasomotor Symptoms (Hot Flashes) From Baseline
Description: Frequency is the number of vasomotor symptoms (hot flashes) recorded by the subject in the continuous diary.
  Week 1
Time Frame: At Week 1 relative to Baseline
Population: Modified intent to treat population included all subjects in the safety population who had at least1 baseline and postbaseline result for an vasomotor symptom parameter. All patients were included. A negative change indicates a reduction.
Measure: Least Squares Mean (Standard Error); unit: hot flashes
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
hot flashes | -2.58 (0.917) | -2.81 (0.918) | -3.60 (0.940) | -3.39 (0.898)

40. Secondary Outcome: Change in Frequency Vasomotor Symptoms (Hot Flashes) From Baseline
Description: Frequency is the number of vasomotor symptoms (hot flashes) recorded by the subject in the continuous diary.
  Week 2
Time Frame: At Week 2 relative to Baseline
Population: as for outcome 39
Measure: Least Squares Mean (Standard Error); unit: hot flashes
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
hot flashes | -3.30 (0.947) | -5.02 (0.948) | -5.15 (0.970) | -5.62 (0.927)

41. Secondary Outcome: Change in Severity of Vasomotor Symptoms (Hot Flashes) From Baseline
Description: Patients recorded in a continuous diary the number of individual hot flashes experienced and rated the severity of each on a scale of mild, moderate, or severe where mild is assigned a value of 1, moderate a value of 2, and severe a value of 3 during data analysis.
  Daily severity was calculated as [(1 × number of mild hot flashes) + (2 × number of moderate hot flashes) + (3 × number of severe hot flashes)]/total number of hot flashes reported. The value at Week 1 was subtracted from the value at Baseline to yield the impact on severity score. A negative change indicates a reduction in severity.
Time Frame: At Week 1 relative to Baseline
Population: Modified intent to treat population included all subjects in the safety population who had at least1 baseline and postbaseline result for an vasomotor symptom parameter. All patients were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
score on a scale | -0.20 (0.067) | -0.20 (0.067) | -0.24 (0.067) | -0.26 (0.065)

42. Secondary Outcome: Change in Severity of Vasomotor Symptoms (Hot Flashes) From Baseline
Description: Patients recorded in a continuous diary the number of individual hot flashes experienced and rated the severity of each on a scale of mild, moderate, or severe where mild is assigned a value of 1, moderate a value of 2, and severe a value of 3 during data analysis.
  Daily severity was calculated as [(1 × number of mild hot flashes) + (2 × number of moderate hot flashes) + (3 × number of severe hot flashes)]/total number of hot flashes reported. The value at Week 2 was subtracted from the value at Baseline to yield the impact on severity score. A negative change indicates a reduction.
Time Frame: At Week 2 relative to Baseline
Population: as for outcome 41
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
score on a scale | -0.31 (0.091) | -0.32 (0.091) | -0.43 (0.091) | -0.37 (0.088)

43. Secondary Outcome: Change in Hot Flash Severity Score Vasomotor Symptoms From Baseline
Description: The hot flash severity score is a composite of the frequency and severity of hot flashes, and was calculated as follows: [number of mild hot flashes on Day Y x 1] + [number of moderate hot flashes on Day Y x 2] + [number of severe hot flashes on Day Y x 3].
  The value at Week 1 was subtracted from the value at Baseline to yield the impact on the composite hot flash severity score. A negative change indicates a reduction.
Time Frame: At Week 1 relative to Baseline
Population: as for outcome 41
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
score on a scale | -6.09 (2.094) | -7.45 (2.082) | -8.10 (2.110) | -8.56 (2.043)

44. Secondary Outcome: Change in Hot Flash Severity Score of Vasomotor Symptoms From Baseline
Description: The hot flash severity score is a composite of the frequency and severity of hot flashes, and was calculated as follows: [number of mild hot flashes on Day Y x 1] + [number of moderate hot flashes on Day Y x 2] + [number of severe hot flashes on Day Y x 3].
  The value at Week 2 was subtracted from the value at Baseline to yield the impact on hot flash severity score. A negative change indicates a reduction in severity.
Time Frame: At Week 2 relative to Baseline
Population: as for outcome 41
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 13
score on a scale | -7.52 (2.214) | -12.47 (2.200) | -11.95 (2.231) | -13.67 (2.159)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- ACER-801 200 mg BID: ACER-801 (osanetant) 200 mg BID (3 x 50 mg and 1 x placebo, twice daily)
  ACER-801 200 mg BID: 200 mg BID (twice daily)
Arm/Group | ACER-801 50 mg BID | ACER-801 100 mg BID | ACER-801 200 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/12 | 0/13
Other Adverse Events (participants affected / at risk) | 9/12 | 7/12 | 6/12 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACER-801 50 mg BID (N=12) | ACER-801 100 mg BID (N=12) | ACER-801 200 mg BID (N=12) | Placebo (N=13)
ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACER-801 50 mg BID (N=12) | ACER-801 100 mg BID (N=12) | ACER-801 200 mg BID (N=12) | Placebo (N=13)
Vessel puncture site pain (General disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Medical device site reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
infusion site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sensation of foreign body (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
vessel puncture site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
frequent bowl movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
vessel puncture site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT05325775/Prot_SAP_001.pdf